CLINICAL TRIAL: NCT04505150
Title: Lowering Blood Pressure by Changing Lifestyle Through a Motivational Education Program: a Cluster RCT Study Protocol
Brief Title: Lowering Blood Pressure by Changing Lifestyle
Acronym: LBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Organisation for Rural Community Development, Bangladesh (Other)
Collaborators: Swinburne University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LBP2723
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: High Blood Pressure
Keywords: lifestyle; health literacy; cluster RCT; physical exercise; smoking
MeSH Terms: conditions — Hypertension; Motor Activity; Smoking

STUDY DESIGN:
Intervention Model Description: Cluster randomised
Masking Description: The individual participant will not be randomly assigned but as a group of participants (intervention arm and control arm) will be randomly selected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring of lifestyle change activities (Experimental): The intervention arm will involve (i) the delivery of a blended learning education program and (ii) weekly phone calls to participants. The lectures will be delivered to 10 teams, comprised of about 15 participants in each team and lead by a volunteer team leader using the ORCD's laptop, overhead projector and the sound system in local clubs, school premises or participants' houses. The ORCD investigator including the physician and an information technology person will facilitate the education programs. The interpretations or additional explanations will be made by the physician following WHO guidelines and recommendations[36]. The investigator will maintain a folder for each team and will communicate at least with the team leaders by phone calls once every week to remind them to adhere to lifestyle modification intervention program. The weekly monitoring program will continue until the study ends.
  Interventions: Behavioral: Lifestyle changes, e.g., take part in regular exercise, quitting smoking, and reduce salt consumption
- lifestyle change activities: non-monitoring (No Intervention): The control group will only receive the printed materials, no active monitoring

INTERVENTIONS:
Behavioral: Lifestyle changes, e.g., take part in regular exercise, quitting smoking, and reduce salt consumption — Intervention participants will receive ongoing counselling with evidence-based information with pictures, fact sheets, published literature about the harmful effect of smoking on hypertension and other cardiovascular diseases for the cessation of smoking and to take part in regular exercise.
  Other Names: Monitoring of lifestyle change activities
  Arms: Monitoring of lifestyle change activities

SUMMARY:
Introduction: High blood pressure is an independent risk factor of cardiovascular disease (CVD) and is a major cause of disability and death. Managing a healthy lifestyle has been shown to reduce blood pressure and improve health outcomes. We aim to investigate the effectiveness of a lifestyle modification intervention program for lowering blood pressure in a rural area of Bangladesh.

Methods and analysis: A single-centre cluster randomized controlled trial (RCT). The study will be conducted for six months, a total of 300 participants of age 30 to 75 years with 150 adults in each of the intervention and the control arms. The intervention arm will involve the delivery of a blended learning education program on lifestyle changes for the management of high blood pressure. The education program comprises evidence-based information with pictures, fact sheets, and published literature about the effects of high blood pressure on CVD development, increased physical activity and the role of a healthy diet in blood pressure management. The control group involves providing information booklets and general advice at the baseline data collection point. The primary outcome will be the absolute difference in clinic systolic and diastolic blood pressure. Secondary outcomes include the difference in the percentage of people adopting regular exercise habits, cessation of smoking and reducing sodium chloride intake, health literacy of all participants, the perceived barriers and enablers to adopt behaviour changes by collecting qualitative data. Analyses will include analysis of covariance to report the mean difference in blood pressure between the control and the intervention group and the difference in change in blood pressure due to the intervention.

DETAILED DESCRIPTION:
High blood pressure is a fundamental cause of cardiovascular disease (CVD) and a major cause of disability and death. Raised blood pressure accounts for as many as 10.4 million deaths per year globally. The prevalence of high blood pressure has increased from 87.0 million in 1999-2000 to 108.2 million in 2015-2016. Of the 1.5 million worldwide annual deaths, 9.4% has been attributed to high blood pressure. Modifiable risk factors such as smoking, unhealthy diet and physical inactivity are shared and established risk factors for CVDs. Lifestyle changes such as smoking cessation, diet alteration including a reduction in dietary sodium intake and increased physical activity can improve health outcomes by decreasing or slowing complications associated with high blood pressure and other CVDs.

Development and subsequent evaluation of effectiveness for any intervention targeting high blood pressure should include core components comprising baseline participant assessment, educational interventions for participants to acquire adequate knowledge about the etiology and risk factors of hypertension, and modification of lifestyle factors such as participating in regular physical activity, consuming a healthy diet and smoking cessation. Despite the high prevalence of high blood pressure in low-income and middle-income countries, there are relatively few data on intervention programs from low-income and middle-income countries (LMICs). Studies also report that a significant proportion of people with high blood pressure are undiagnosed or do not meet targets to control blood pressure both in developed and in LMICs. Among people with known high blood pressure, less than one-third of people are able to control their high blood pressure with appropriate treatment. Lifestyle modification programs have been shown to be effective in controlling blood pressure in LMICs.

Bangladesh, a low-income country in South East Asia, is currently confronting an increasing burden of chronic diseases, including high blood pressure. Islam et al. conducted a cross-sectional study among adults age ≥30 years in a rural district in Bangladesh that reported the knowledge, attitudes and practice of diabetes and common eye diseases, and found overall knowledge was below average. The study also reported the prevalence and risk factors associated with known and undiagnosed diabetes, and self-reported known high blood pressure and newly diagnosed high blood pressure. The study identified that 40% of adults had high blood pressure, of which 82% were previously undiagnosed. Almost 60% of those with high blood pressure also had diabetes.

Recently, a community-based cluster randomized controlled trial was conducted in rural communities in Bangladesh, Pakistan and Sri Lanka. This multicomponent intervention program was conducted for 24 months in 2645 adults with hypertension defined as blood pressure greater than or equal to 140/90 mm Hg. The study reported a statistically significant mean reduction of systolic blood pressure of 5.2 mm Hg from the baseline mean blood pressure 146.7 mm Hg compared to the usual care in which the reduction was 3.9 mm Hg. Relatively small reductions of 2 mm Hg in SBP and DBP have been reported to lower the risk of stroke by 14% and 17%, respectively, and the risk of coronary artery disease by 9% and 6%, respectively. The intervention program included home visits by government community health workers for blood-pressure monitoring and counselling and the training of physicians. A possible limitation of this intervention program maybe that home visits by trained community health workers for blood pressure monitoring and counselling may not be a sustainable and cost-saving approach due to the shortage of qualified workforce and the budget constraints in low- middle-income countries. Application of blended learning education programs to educate patients in managing blood pressure by changing lifestyle and participation in intervention programs as volunteers coordinated by volunteer leaders may be a sustainable approach for lowering blood pressure in the community setting. The goal of this pilot study is to compare a multicomponent intervention program to evaluate its effectiveness for lowering blood pressure among adults with high blood pressure in a rural district in Bangladesh.

Health literacy is a complex and combined perception comprising a range of attributes including available resources of health-related information, and an individuals' intellectual, emotional, social and personal skills. Health literacy empowers people with skills to improve their health and well-being. Evidence indicates that deficits in health literacy are associated with poorer health outcomes and higher health-related costs at both individual and system levels. Improved health literacy had been reported to be associated with reductions in risk behaviours for chronic disease. However, an extended and often asymptomatic onset and a need for ongoing management, these conditions present people with a sharp and upward learning curve about risks, treatments and self-care. Self-care, especially in resource-limited settings, an essential dimension of treatment, depends on the ability of systems and providers to teach and patients to learn effective self-management skills. At the individual level, good health literacy is the foundation of successful management and prevention of chronic disease. Health literacy assessment can be used to improve community participation in health, health service planning, public health education, and policy development. In the past decade, much research on the impact of health literacy on health outcomes has been conducted across the globe; however, health literacy tools in rural areas of Bangladesh have not been developed or tested. The European Health Literacy Survey (HLS- Q12) questionnaire has been used to assess health literacy; however, its usefulness to measure health literacy in rural Bangladesh has not been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Participants with clinic blood pressure more than or equal to 130/80 mm Hg who are not taking medication
* Participants with controlled blood pressure defined as < 130/80 using anti-hypertensive medication for a minimum of six weeks.
* Participants live in Banshgram Union only

Exclusion Criteria:

* Aged > 75 years of age
* Pregnant women
* People who have advanced CVDs or are any serious condition that restricts their participation in the study
* Participants will be withdrawn from the study if they are unwilling to continue their participation and withdraw their consent, or any women participants who become pregnant during the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure in mmHg | 1. Baseline, 2. during the intervention (3 months) and 3. Immediately after the intervention (six months)
  Data at baselie will be compared between the control and intervention arms; change will be computed from the difference between three and six months from baseline measures and will be compared between and within groups. Omron blood pressure measuring tool will be used.

SECONDARY OUTCOMES:
Evaluation of the psychometric properties of a Health literacy tool, European Health Literacy Survey Questionnaire (HLS-Q12) in rural Bangladesh. | Baseline
  Psychometric properties of a Health literacy tool will be investigated. HLQ12 is a 12 item questionnaire developed to measure health literacy related to knowledge of and access to health. The Questionnaire was developed and valided in European countries but it is not known whether all items are appropriate in any developing countries such as in Bangladesh. Therefore, using Rasch analysis, we could investigate if 12 items are necessary or need any modifications. Therefore, the outcome measure is the tool itself. Do we need all the items or not?
Assesment of the level of health literacy using health related scale European Health Literacy Survey Questionnaire | 1. Baseline and 2. Immediately after the intervention (six months)
  Estimate the current level of health literacy. After assessing psychometric properties, we may come up with all 12 or removing one or two items. Based on these items, we will be able to report the proportion of people who have a higher/lower level of health literacy. For example, 70 percent of people with higher education are able to access to health facilities, can read prescriptions or can take a decision which physicians they need to go compared to 30 per cent in people who are illiterate. Outcome: proportion. Each item of the scale has four categories (1-4), 1 is associated low level of literacy and 4 mean high level of literacy
Barriers and enablers in managing healthy lifestyle in a rural area in Bangladesh | 1. Immediately after the intervention (six months)
  Qualitative data will be collected from 10 participants and five health professionals and study coordinator. This is qualitative information from the participants to investigate the perceived barriers and enablers to scale up this study. The software NVivo will be used to investigate if there are any common themes of barriers which could intervene. This is descriptive information.
Mobile use, reading SMS, intention to receive SMS for health information in people with high blood pressure in a rural area in Bangladesh | 1. Baseline
  percentage of people who owns a mobile, can read SMS and willing to receive SMS and pay for it. Outcomes: Proportion
Physical activity levels and intention to take part in physical activities in people with high blood pressure: A cluster RCT | 1. Baseline and 2. Immediately after the intervention (six months)
  Physical activity levels and their correlation with the socio-demographic factors (reported as proporion and relative risk), and intention to take part in physical activity program (reported as proporion and relative risk) in people with high blood pressure in a rural area in Bangladesh. Tool: Global Physical Activity Questionnaire (GPAQ). There are 17 items with "yes" and "no" responses. Yes indicates people take part in physical activity and "no" means they do not take part in physical activity.
Tobacco smoking and use of smokeless tobacco, and intention to quit among people with high blood pressure in a rural area in Bangladesh | 1. Baseline and 2. Immediately after the intervention (six months)
  Proportion of people who smoke tobacco and consume smokeless tobacco. What are the proportion of people who intend to quit smoking or reduce smoking within next three months or six months, and associated socio-demographic factors. Tool: Smoking cessation motivation questionnaire (Q-MAT). The Q-MAT has 19 items. Some items have "yes" and "no" responses and some items have 1-5 scores such as item 4: Do you think that smoking is bad for your health with possible responses are: 1.Not at all 2. A little 3. A lot 4. Enormously 5. I do not know.
Perception of and practice in salt and fruit consumptions and their associations with high blood pressure | 1. Baseline and 3. Immediately after the intervention (six months)
  Proportion of people who are aware that raw salt is not good for blood pressure, what are the factors associated, who are aware of healthy diet and how many people have been practicing. Tool: A modified version of Q-MAT

CONTACTS AND LOCATIONS:
Overall Officials: Fakir M Amirul Islam, PhD, Principal Investigator — Organisation for Rural Community Development
Locations (1):
- Organisation for Rural Community Development, Narail, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other researchers for collaborations
Supporting Information: Study Protocol, SAP
Time Frame: After two years of data collection
Access Criteria: Contact with the chief investigator: amirul.islam@orcdbd.org; fislam@swin.edu.au
URL: http://www.orcdbd.org

REFERENCES:
- [Background] GBD 2017 Risk Factor Collaborators. Global, regional, and national comparative risk assessment of 84 behavioural, environmental and occupational, and metabolic risks or clusters of risks for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1923-1994. doi: 10.1016/S0140-6736(18)32225-6. Epub 2018 Nov 8. PMID 30496105
- [Background] Boehme AK, Esenwa C, Elkind MS. Stroke Risk Factors, Genetics, and Prevention. Circ Res. 2017 Feb 3;120(3):472-495. doi: 10.1161/CIRCRESAHA.116.308398. PMID 28154098
- [Background] Mills KT, Bundy JD, Kelly TN, Reed JE, Kearney PM, Reynolds K, Chen J, He J. Global Disparities of Hypertension Prevalence and Control: A Systematic Analysis of Population-Based Studies From 90 Countries. Circulation. 2016 Aug 9;134(6):441-50. doi: 10.1161/CIRCULATIONAHA.115.018912. PMID 27502908
- [Background] Islam FM, Bhuiyan A, Chakrabarti R, Rahman MA, Kanagasingam Y, Hiller JE. Undiagnosed hypertension in a rural district in Bangladesh: The Bangladesh Population-based Diabetes and Eye Study (BPDES). J Hum Hypertens. 2016 Apr;30(4):252-9. doi: 10.1038/jhh.2015.65. Epub 2015 Jun 25. PMID 26108363
- [Background] Dorans KS, Mills KT, Liu Y, He J. Trends in Prevalence and Control of Hypertension According to the 2017 American College of Cardiology/American Heart Association (ACC/AHA) Guideline. J Am Heart Assoc. 2018 Jun 1;7(11):e008888. doi: 10.1161/JAHA.118.008888. PMID 29858369
- [Background] Carey RM, Muntner P, Bosworth HB, Whelton PK. Prevention and Control of Hypertension: JACC Health Promotion Series. J Am Coll Cardiol. 2018 Sep 11;72(11):1278-1293. doi: 10.1016/j.jacc.2018.07.008. PMID 30190007
- [Background] Halcomb E, Moujalli S, Griffiths R, Davidson P. Effectiveness of general practice nurse interventions in cardiac risk factor reduction among adults. JBI Libr Syst Rev. 2007;5(7):407-453. doi: 10.11124/01938924-200705070-00001. PMID 27820062
- [Background] Balady GJ, Williams MA, Ades PA, Bittner V, Comoss P, Foody JA, Franklin B, Sanderson B, Southard D; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee; Council on Clinical Cardiology; Councils on Cardiovascular Nursing, Epidemiology and Prevention, and Nutrition, Physical Activity, and Metabolism; American Association of Cardiovascular and Pulmonary Rehabilitation. Core components of cardiac rehabilitation/secondary prevention programs: 2007 update: a scientific statement from the American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee, the Council on Clinical Cardiology; the Councils on Cardiovascular Nursing, Epidemiology and Prevention, and Nutrition, Physical Activity, and Metabolism; and the American Association of Cardiovascular and Pulmonary Rehabilitation. J Cardiopulm Rehabil Prev. 2007 May-Jun;27(3):121-9. doi: 10.1097/01.HCR.0000270696.01635.aa. PMID 17558191
- [Background] Rehabilitation after cardiovascular diseases, with special emphasis on developing countries. Report of a WHO Expert Committee. World Health Organ Tech Rep Ser. 1993;831:1-122. No abstract available. PMID 8351937
- [Background] Grace SL, Turk-Adawi KI, Contractor A, Atrey A, Campbell N, Derman W, Melo Ghisi GL, Oldridge N, Sarkar BK, Yeo TJ, Lopez-Jimenez F, Mendis S, Oh P, Hu D, Sarrafzadegan N. Cardiac rehabilitation delivery model for low-resource settings. Heart. 2016 Sep 15;102(18):1449-55. doi: 10.1136/heartjnl-2015-309209. Epub 2016 May 15. PMID 27181874
- [Background] Head GA, Shaw JE, Dunstan DW, Owen N, Magliano DJ, Chadban S, Zimmet P. Hypertension, white-coat hypertension and masked hypertension in Australia: findings from the Australian Diabetes, Obesity, and Lifestyle Study 3. J Hypertens. 2019 Aug;37(8):1615-1623. doi: 10.1097/HJH.0000000000002087. PMID 31058796
- [Background] Arokiasamy P, Uttamacharya, Kowal P, Capistrant BD, Gildner TE, Thiele E, Biritwum RB, Yawson AE, Mensah G, Maximova T, Wu F, Guo Y, Zheng Y, Kalula SZ, Salinas Rodriguez A, Manrique Espinoza B, Liebert MA, Eick G, Sterner KN, Barrett TM, Duedu K, Gonzales E, Ng N, Negin J, Jiang Y, Byles J, Madurai SL, Minicuci N, Snodgrass JJ, Naidoo N, Chatterji S. Chronic Noncommunicable Diseases in 6 Low- and Middle-Income Countries: Findings From Wave 1 of the World Health Organization's Study on Global Ageing and Adult Health (SAGE). Am J Epidemiol. 2017 Mar 15;185(6):414-428. doi: 10.1093/aje/kww125. PMID 28399566
- [Background] Geldsetzer P, Manne-Goehler J, Marcus ME, Ebert C, Zhumadilov Z, Wesseh CS, Tsabedze L, Supiyev A, Sturua L, Bahendeka SK, Sibai AM, Quesnel-Crooks S, Norov B, Mwangi KJ, Mwalim O, Wong-McClure R, Mayige MT, Martins JS, Lunet N, Labadarios D, Karki KB, Kagaruki GB, Jorgensen JMA, Hwalla NC, Houinato D, Houehanou C, Msaidie M, Guwatudde D, Gurung MS, Gathecha G, Dorobantu M, Damasceno A, Bovet P, Bicaba BW, Aryal KK, Andall-Brereton G, Agoudavi K, Stokes A, Davies JI, Barnighausen T, Atun R, Vollmer S, Jaacks LM. The state of hypertension care in 44 low-income and middle-income countries: a cross-sectional study of nationally representative individual-level data from 1.1 million adults. Lancet. 2019 Aug 24;394(10199):652-662. doi: 10.1016/S0140-6736(19)30955-9. Epub 2019 Jul 18. PMID 31327566
- [Background] Yusuf S, Joseph P, Rangarajan S, Islam S, Mente A, Hystad P, Brauer M, Kutty VR, Gupta R, Wielgosz A, AlHabib KF, Dans A, Lopez-Jaramillo P, Avezum A, Lanas F, Oguz A, Kruger IM, Diaz R, Yusoff K, Mony P, Chifamba J, Yeates K, Kelishadi R, Yusufali A, Khatib R, Rahman O, Zatonska K, Iqbal R, Wei L, Bo H, Rosengren A, Kaur M, Mohan V, Lear SA, Teo KK, Leong D, O'Donnell M, McKee M, Dagenais G. Modifiable risk factors, cardiovascular disease, and mortality in 155 722 individuals from 21 high-income, middle-income, and low-income countries (PURE): a prospective cohort study. Lancet. 2020 Mar 7;395(10226):795-808. doi: 10.1016/S0140-6736(19)32008-2. Epub 2019 Sep 3. PMID 31492503
- [Background] Jafar TH, Gandhi M, de Silva HA, Jehan I, Naheed A, Finkelstein EA, Turner EL, Morisky D, Kasturiratne A, Khan AH, Clemens JD, Ebrahim S, Assam PN, Feng L; COBRA-BPS Study Group. A Community-Based Intervention for Managing Hypertension in Rural South Asia. N Engl J Med. 2020 Feb 20;382(8):717-726. doi: 10.1056/NEJMoa1911965. PMID 32074419
- [Background] Saquib N, Saquib J, Ahmed T, Khanam MA, Cullen MR. Cardiovascular diseases and type 2 diabetes in Bangladesh: a systematic review and meta-analysis of studies between 1995 and 2010. BMC Public Health. 2012 Jun 13;12:434. doi: 10.1186/1471-2458-12-434. PMID 22694854
- [Background] Islam FM, Chakrabarti R, Dirani M, Islam MT, Ormsby G, Wahab M, Critchley C, Finger RP. Knowledge, attitudes and practice of diabetes in rural Bangladesh: the Bangladesh Population based Diabetes and Eye Study (BPDES). PLoS One. 2014 Oct 14;9(10):e110368. doi: 10.1371/journal.pone.0110368. eCollection 2014. PMID 25313643
- [Background] Islam FM, Chakrabarti R, Islam SZ, Finger RP, Critchley C. Factors Associated with Awareness, Attitudes and Practices Regarding Common Eye Diseases in the General Population in a Rural District in Bangladesh: The Bangladesh Population-based Diabetes and Eye Study (BPDES). PLoS One. 2015 Jul 22;10(7):e0133043. doi: 10.1371/journal.pone.0133043. eCollection 2015. PMID 26200458
- [Background] Islam FM, Chakrabarti R, Islam MT, Wahab M, Lamoureux E, Finger RP, Shaw JE. Prediabetes, diagnosed and undiagnosed diabetes, their risk factors and association with knowledge of diabetes in rural Bangladesh: The Bangladesh Population-based Diabetes and Eye Study. J Diabetes. 2016 Mar;8(2):260-8. doi: 10.1111/1753-0407.12294. Epub 2015 May 6. PMID 25851830
- [Background] Finbraten HS, Wilde-Larsson B, Nordstrom G, Pettersen KS, Trollvik A, Guttersrud O. Establishing the HLS-Q12 short version of the European Health Literacy Survey Questionnaire: latent trait analyses applying Rasch modelling and confirmatory factor analysis. BMC Health Serv Res. 2018 Jun 28;18(1):506. doi: 10.1186/s12913-018-3275-7. PMID 29954382
- [Background] Dansou A, Groussin L, Gaborit C, Touraine A, Blanchet E, Laporte L, Jouneau C, Pennamen E, Maino B. [Approach and management of tobacco quitting process of the smoker patient by 149 residents in a university hospital in Tours]. Rev Mal Respir. 2012 Sep;29(7):878-88. doi: 10.1016/j.rmr.2012.02.010. Epub 2012 Jun 6. French. PMID 22980548
- [Background] Mumu SJ, Ali L, Barnett A, Merom D. Validity of the global physical activity questionnaire (GPAQ) in Bangladesh. BMC Public Health. 2017 Aug 10;17(1):650. doi: 10.1186/s12889-017-4666-0. PMID 28797237
- [Background] Chu AH, Ng SH, Koh D, Muller-Riemenschneider F. Reliability and Validity of the Self- and Interviewer-Administered Versions of the Global Physical Activity Questionnaire (GPAQ). PLoS One. 2015 Sep 1;10(9):e0136944. doi: 10.1371/journal.pone.0136944. eCollection 2015. PMID 26327457
- [Derived] Amirul Islam FM. Study of the psychometric properties of the HLS-EU-12 questionnaire in rural Bangladesh. PLoS One. 2025 May 12;20(5):e0323608. doi: 10.1371/journal.pone.0323608. eCollection 2025. PMID 40354386
- [Derived] Islam FMA, Lambert EA, Islam SMS, Islam MA, Biswas D, McDonald R, Maddison R, Thompson B, Lambert GW. Lowering blood pressure by changing lifestyle through a motivational education program: a cluster randomized controlled trial study protocol. Trials. 2021 Jul 8;22(1):438. doi: 10.1186/s13063-021-05379-2. PMID 34238363